CLINICAL TRIAL: NCT02411864
Title: Can the Distribution of Low B-value and the NEX Influence the Pseudodiffusion Parameter Derived From IVIM in Brain?
Brief Title: Optimal Low B-value in Intravoxel Incoherent Motion Diffusion-weighted MR Imaging of the Brain
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDLL-20140570
Record Dates: First submitted 2014-12-10; First posted 2015-04-08 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteers
Keywords: IVIM; brain; diffusion-weighted imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group 1: Low b=(0,50,150,200)，NEX=(1,3,2,2)
  Interventions: Other: different low b-values distribution
- Group 2: Low b=(0,30,50,100,200)，NEX=(1,3,3,2,2)
  Interventions: Other: different low b-values distribution
- Group 3: Low b=(0,30,60,90,120,150,180,200)，NEX=(1,3,3,3,2,2,2,2)
  Interventions: Other: different low b-values distribution
- Group 4: Low b=(0,30,60,90,120,150,180,200)，NEX=(1,1,1,1,1,1,1,1)
- Group 5: Low b=(0,20,40,60,80,100,120,140,160,180,200)NEX=(1,3,3,3,3,2,2
  Interventions: Other: different low b-values distribution

INTERVENTIONS:
Other: different low b-values distribution
  Groups: Group 1; Group 2; Group 3; Group 5

SUMMARY:
Our research aims to reveal whether the low b-values distribution and the number of NEX for each b value will influence the accuracy of pseudodiffusion parameter derived from IVIM in brain.

DETAILED DESCRIPTION:
As an improved MRI technique, diffusion-weighted imaging (DWI) is considered the most sensitive for early pathological changes. Perfusion measurement has been shown to improve sensitivity and predictive value for tumor grading and prognosis, also as a predicator of recovery with reperfusion in patients of acute ischemic stroke.Our research aims to reveal whether the low b-values distribution and the number of NEX for each b value will influence the accuracy of pseudodiffusion parameter derived from IVIM in brain.

ELIGIBILITY:
Inclusion Criteria:

* no hypertension or cerebral vascular diseases,
* no systemic metabolic disease;
* no infection or fever;
* no use of corticosteroid drugs;
* no MRI contraindication.

Exclusion Criteria:

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Parameters D* and f in healthy white matter or gray mater | 2-3 days